CLINICAL TRIAL: NCT01060722
Title: A Phase I, Randomized, Double-Blinded, Placebo-Controlled, Single-Dose, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of a Long Acting Human Growth Hormone (hGH) Product (MOD-4023), in Healthy Volunteers
Brief Title: MOD-4023 Study in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Collaborators: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CP-4-001
Record Dates: First submitted 2010-01-31; First posted 2010-02-02 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Healthy
Keywords: Healthy Male Volunteers
MeSH Terms: interventions — MOD-4023

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- MOD-4023, dose level 1 (Experimental)
  Interventions: Drug: MOD-4023 (long lasting hGH); Drug: Placebo
- MOD-4023, dose level 2 (Experimental)
  Interventions: Drug: MOD-4023 (long lasting hGH); Drug: Placebo
- MOD-4023, dose level 3 (Experimental)
  Interventions: Drug: MOD-4023 (long lasting hGH); Drug: Placebo

INTERVENTIONS:
Drug: MOD-4023 (long lasting hGH) — Single subcutaneous dose of MOD-4023
Drug: Placebo — Single subcutaneous dose of placebo material

SUMMARY:
This study aims to examine the safety, tolerability and pharmacokinetics of a long-lasting Human Growth Hormone (MOD-4023) in healthy volunteers after a single subcutaneous injection at escalating doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers aged 18-45 (inclusive) years.
* Body Mass Index (BMI) 19 to 30 kg/m2 (inclusive) and weighing at least 55 Kg.
* Non-smoking (by declaration) for a period of at least 6 months prior to screening visit.
* Subjects in generally good health in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
* Blood pressure and heart rate within normal limits (blood pressure: systolic 90-140mmHg; diastolic 50-90 mmHg, heart rate 40-100 beats per minute).
* Electrocardiogram (ECG) with no clinically significant abnormalities recorded at screening visit (up to 21 days before dosing) and on dosing day (before drug administration): PR interval within 120 and 200 ms, QRS interval < 120 ms, and QTc interval ≤ 440 ms.
* Negative HIV, hepatitis B or hepatitis C serology tests at screening
* No clinically significant abnormalities in complete blood count (CBC), prothrombin time (PT, INR), activated partial thromboplastin time (aPTT), chemistry lab tests (liver and renal function) and urinalysis at screening.
* No history of alcohol or drug abuse. Negative urine DoA in screening and on admission. Negative breath alcohol on admission.
* Subjects must agree to use medically accepted form of contraception from dosing day to 12 weeks after drug administration.
* Subjects must be able to understand the requirements of the study and must be willing to comply with the requirements of the study and to provide their written informed consent to participate in the study.

Exclusion Criteria:

* History of significant neurological (including history of seizures or EEG abnormalities), renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrinological, gastrointestinal, hematopoietic disease, neoplasm, psychological (marked anxiety, tension or agitation) or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medication.
* Diabetes.
* Known allergy to any drug.
* Adherence (for whatever reason) to an abnormal diet during the 4 weeks prior to the study, or subjects with recent significant change in body weight.
* Use of any prescription or over-the-counter (OTC) medications, including vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
* Subjects who have received any vaccines within 4 weeks prior to study drug administration.
* Subjects who donated blood in the three months or received blood or plasma derivatives in the six months preceding study drug administration.
* Participation in another clinical trial with drugs within 3 months prior to dosing (calculated from the previous study's last dosing date).
* Subjects with an inability to communicate well with the investigators and CRC staff (i.e., language problem, poor mental development or impaired cerebral function).
* Subjects that have difficulty fasting or consuming the standard meals that will be provided.
* Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
* Subjects who are non-cooperative or unwilling to sign a consent form.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability (AE's, vital signs, ECG, laboratory tests, local reaction) | 30 days
Pharmacokinetics: AUC, Cmax, Tmax, T1/2 | 14 days

SECONDARY OUTCOMES:
Formation of anti-drug antibodies | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Atsmon, M.D., Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel